CLINICAL TRIAL: NCT02987725
Title: Laboratory-based Hypnosis Intervention on Pain Responsivity in Adolescents With Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sarah R. Martin, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: F32sarahmartin2
Record Dates: First submitted 2016-12-01; First posted 2016-12-09 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Sickle Cell Disease
Keywords: Adolescence; Autonomic Nervous System; Hypnosis; Pain; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell; Pain | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Control (Active Comparator): Participants will listen to a 30-minute historical story.
  Interventions: Behavioral: Attention Control
- Hypnosis (Experimental): Participants will receive a 30-minute hypnosis session
  Interventions: Behavioral: Hypnosis

INTERVENTIONS:
Behavioral: Hypnosis — A 30-minute Hypnosis session with a trained clinician focused on relaxation and hypnotic suggestions for pain relief and reduced stress responses.
  Arms: Hypnosis
Behavioral: Attention Control — A 30-minute historical story read by a research clinician.
  Arms: Attention Control

SUMMARY:
The purpose of this study is to test the effects of a laboratory-based hypnosis session compared to an attention control condition on peripheral blood flow, autonomic stress responses, and acute pain responses in adolescents (ages 12-21) with sickle cell disease, and examine how perceived disease-related stigma may affect these responses.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of sickle cell disease
* Age 12-21 years old
* Fluent in English (the intervention will be delivered in English)
* Participant is cognitively able to provide informed signed consent or assent
* Participant is cognitively able to follow instructions

Exclusion Criteria:

* Under 12 years of age or over 21 years of age
* Not fluent in English
* Pain medication prescription has changed or if they have been hospitalized for a vaso-occlusive episode within 30 days of study participation.
* Diagnosis of a condition (e.g., neurological disorder affecting peripheral sensation, skin abnormality over the stimulus site, obstructive sleep apnea, diabetes, ischemic heart disease) or cognitive impairment that may affect data integrity or the ability to complete study procedures.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Change in peripheral blood flow before and during the intervention | Beginning 15 minutes prior to the intervention (hypnosis or attention control) and continuing during 30 minutes of the intervention
  Peripheral blood flow will be measured using continuous readings of oxygen saturation, pulse rate, and pulse waveform from the thumb and change in blood flow will be assessed by comparing levels of blood flow during the pre-intervention period (15 minutes prior to intervention to a minute before the start of intervention) from blood flow during the intervention period (from the start of the intervention until 30 minutes after the start of the intervention).

SECONDARY OUTCOMES:
Change in pain threshold temperature | 12 minutes before the start of the intervention and 15 minutes after the start of the intervention.
  Pain threshold temperature will be determined by when participants report they first feel pain and change in pain threshold temperature will be assessed by comparing pain threshold temperature during the pre-intervention period (12 minutes before the start of the intervention) from pain threshold temperature during the intervention period (15 minutes after the start of the intervention).
Change in pain tolerance temperature | 9 minutes before the start of the intervention and 18 minutes after the start of the intervention.
  Pain tolerance temperature will be determined by when participants report they can no longer tolerate the pain and change in pain tolerance temperature will be assessed by comparing pain tolerance temperature during the pre-intervention period (9 minutes before the start of the intervention) from pain tolerance temperature during the intervention period (18 minutes after the start of the intervention).
Change in heat pulse pain intensity ratings | 5 minutes before the start of the intervention and 21 minutes after the start of the intervention.
  Heat pulse pain intensity ratings will be determined by participants' self-report of heat pulse pain intensity (rated on a 0-10 scale, with 0 being no pain and 10 being worst pain), and change in heat pulse pain intensity will be assessed by comparing pain tolerance temperature during the pre-intervention period (5 minutes before the start of the intervention) from heat pulse pain intensity during the intervention period (21 minutes after the start of the intervention).
Change in the effect of the intervention on peripheral blood flow at different levels of disease-related stigma | 15 minutes prior to the start of the intervention to a minute before the start of the intervention and from the start of the intervention to 30 minutes after the start of the intervention
  Stigma will be assessed via a questionnaire completed prior to the start of the laboratory session and will be compared to the change in effect, which is assessed by comparing levels of blood flow during the pre-intervention period (15 minutes prior to intervention to a minute before the start of intervention) from blood flow during the intervention period (from the start of the intervention until 30 minutes after the start of the intervention).
Change in the effect of the intervention on pain threshold temperature at different levels of disease-related stigma | 12 minutes before the start of the intervention and 15 minutes after the start of the intervention
  Stigma will be assessed via a questionnaire completed prior to the start of the laboratory session and will be compared to the change in effect, which is assessed by comparing pain threshold collected 12 minutes before the start of the intervention and 15 minutes after the start of the intervention.
Change in the effect of the intervention on pain tolerance temperature at different levels of disease-related stigma | 9 minutes before the start of the intervention and 18 minutes after the start of the intervention.
  Stigma will be assessed via a questionnaire completed prior to the start of the laboratory session and will be compared to the change in effect, which is assessed by comparing pain tolerance collected 9 minutes before the start of the intervention and 18 minutes after the start of the intervention.
Change in the effect of the intervention on heat pulse pain intensity ratings at different levels of disease-related stigma | 5 minutes before the start of the intervention and 21 minutes after the start of the intervention.
  Stigma will be assessed via a questionnaire completed prior to the start of the laboratory session and will be compared to the change in effect, which is assessed by comparing pain intensity collected 5 minutes before the start of the intervention and 21 minutes after the start of the intervention.

OTHER OUTCOMES:
Change in the effect of the intervention on Skin Conductance Response (SCR) | 12-5 minutes prior to the start of the intervention and 15-21 minutes after the start of the intervention
  Skin Conductance Response (SCR) will be measured using continuous readings of electrical properties of the skin on the index finger and change in SCR will be assessed by comparing levels of SCR during the pre-intervention period (12-5 minutes prior to intervention to the start of intervention) from SCR during the intervention period (15-21 minutes after the start of the intervention).
Change in the effect of the intervention on Heart Rate Variability | 12-5 minutes prior to the start of the intervention and 15-21 minutes after the start of the intervention
  Heart Rate Variability (HRV) will be measured using continuous readings of heartbeat intervals and change in HRV will be assessed by comparing HRV during the pre-intervention period (12-5 minutes prior to intervention to the start of intervention) from HRV during the intervention period (15-21 minutes after the start of the intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Lonnie K Zeltzer, MD, Study Chair — UCLA Pediatric Pain and Palliative Care Program
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States